CLINICAL TRIAL: NCT06615518
Title: "Radiological Analysis of MRI Images in Patients Treated With Minimally Invasive Microsurgical and Endoscopic Techniques: A Randomized Study Comparing the Clinical Effectiveness of Full Endoscopic Lumbar Discectomy (FELD) and Microdiscectomy (MD)"
Brief Title: Comparison of Clinical Effectiveness of Full Endoscopic Lumbar Discectomy (FELD) and Microdiscectomy (MD) in Patients With Lumbar Disc Herniation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Opole (Other)
Responsible Party: Principal Investigator, Kajetan Latka, PhD, Deputy-Head Neurosurgery Department WSS Opole, University of Opole
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UO/0001/KB/2024
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Degenerative Disease; Lumbar Radiculopathy; Sciatic Leg Pain; Sciatic Nerve Compression; Discopathy; Disc Herniation; Disc Herniation With Radiculopathy
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TELD (Experimental): Transforaminal endoscopic lumbar discectomy
  Interventions: Procedure: transforaminal endoscopic lumbar discectomy
- IELD (Experimental): Interlaminar endoscopic lumbar discectomy
  Interventions: Procedure: Interlaminar endoscopic lumbar discectomy
- MD (Active Comparator): microdiscectomy
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: transforaminal endoscopic lumbar discectomy — FELD is a minimally invasive spine surgery technique performed through small incisions using an endoscope. The procedure involves accessing the herniated disc through either the transforaminal (TELD) or interlaminar (IELD) approach, depending on the location of the disc herniation. The endoscopic approach allows for direct visualization of the affected area using a camera, and specialized instruments are used to remove the herniated portion of the disc.
  What distinguishes this intervention:
  * Small incisions (typically <1 cm) result in less soft tissue damage compared to traditional open surgery.
  * Real-time endoscopic visualization allows for precise disc removal and reduced trauma to surrounding structures such as muscles and ligaments.
  * Minimized postoperative pain and faster recovery times due to the less invasive nature of the procedure.
  * Outpatient or short hospital stay is often possible, contributing to faster patient discharge.
  Arms: TELD
Procedure: Interlaminar endoscopic lumbar discectomy — FELD is a minimally invasive spine surgery technique performed through small incisions using an endoscope. The procedure involves accessing the herniated disc through either the transforaminal (TELD) or interlaminar (IELD) approach, depending on the location of the disc herniation. The endoscopic approach allows for direct visualization of the affected area using a camera, and specialized instruments are used to remove the herniated portion of the disc.
  What distinguishes this intervention:
  * Small incisions (typically <1 cm) result in less soft tissue damage compared to traditional open surgery.
  * Real-time endoscopic visualization allows for precise disc removal and reduced trauma to surrounding structures such as muscles and ligaments.
  * Minimized postoperative pain and faster recovery times due to the less invasive nature of the procedure.
  * Outpatient or short hospital stay is often possible, contributing to faster patient discharge.
  Arms: IELD
Procedure: Microdiscectomy — Microdiscectomy is a conventional surgical technique for treating lumbar disc herniation, involving a small open incision. In this procedure, the surgeon makes an incision typically between 2-3 cm in length, then uses an operating microscope to gain magnified visualization of the herniated disc. The surgeon removes part of the lamina (laminotomy) to access the disc and nerves. Special instruments are used to remove the herniated portion of the disc that is compressing the spinal nerves, relieving symptoms such as pain, numbness, and weakness.
  What distinguishes this intervention:
  * Larger incision (2-3 cm) compared to FELD, but still smaller than traditional open discectomy, allowing better visualization.
  * Microscopic magnification allows precise removal of disc material while minimizing trauma to surrounding neural structures.
  * Direct access to the affected area via the removal of part of the lamina (laminotomy), offering a well-established and highly effective approach to reli
  Arms: MD

SUMMARY:
The goal of this clinical trial is to compare the clinical effectiveness of Full Endoscopic Lumbar Discectomy (FELD) and Microdiscectomy (MD) in patients aged 18-85 with single-level lumbar disc herniation who have not undergone prior lumbar surgery. This study also aims to perform a radiological analysis of MRI scans before and after treatment to optimize patient selection and surgical strategies. The main questions it aims to answer are:

* Does FELD provide superior early postoperative pain relief (measured by VAS) compared to MD?
* Does FELD offer better functional recovery (measured by COMI and ODI scores) postoperatively compared to MD?
* Can radiological analysis of pre- and post-operative MRI images help optimize patient qualification and guide surgical strategies?

Researchers will compare patients undergoing FELD to those undergoing MD to see if endoscopic techniques result in faster recovery and lower early postoperative pain while maintaining similar long-term outcomes. The study will also analyze how MRI findings correlate with clinical outcomes to refine operative decision-making.

Participants will:

* Undergo either FELD or MD surgery
* Complete VAS, COMI, and ODI questionnaires at pre-specified follow-up intervals (1, 3, 6, and 12 months post-surgery)
* Have MRI scans 24 hours before surgery, 24 hours after surgery, and at each follow-up to assess disc recurrence, residual pathology, and to optimize surgical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years with symptoms of sciatica lasting more than 6 weeks
* Shorter duration in cases where symptoms significantly impair normal functioning or in cases of muscle strength deficits
* Symptoms correlate with MRI findings of lumbar spine pathology, showing the presence of intervertebral disc herniation (protrusion, extrusion, or sequestration) causing nerve root compression in the lumbar spine.

Exclusion Criteria:

* Previous lumbar spine surgery in the lumbar-sacral region
* MRI findings showing degenerative or stenotic spinal canal changes
* Multi-level pathology where identification of the pain source is not possible
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Back and Leg Pain Intensity (measured by the Visual Analog Scale [VAS]) | Baseline, 1 month, 3 months, 6 months, 12 months post-surgery
  Description: The primary outcome measure will assess changes in back and leg pain intensity reported by patients using the Visual Analog Scale (VAS) at each follow-up. The reduction in pain scores will be compared between the FELD and MD groups to evaluate which technique provides superior pain relief over time.

SECONDARY OUTCOMES:
Change in Functional Disability (measured by the Oswestry Disability Index [ODI]) | Baseline, 1 month, 3 months, 6 months, 12 months post-surgery
  This measure will assess the improvement in functional disability using the ODI, comparing the degree of disability reduction between the FELD and MD groups at each follow-up point.
Change in Overall Patient Well-Being (measured by the Core Outcome Measures Index [COMI]) | Baseline, 1 month, 3 months, 6 months, 12 months post-surgery
  The COMI questionnaire will be used to evaluate changes in the patient's overall perception of their condition, including pain, function, and quality of life. Comparisons will be made between FELD and MD groups to assess which method leads to a greater improvement in patient well-being.
Recurrence Rate of Disc Herniation (measured by MRI and clinical assessment) | 1 month, 3 months, 6 months, 12 months post-surgery
  The rate of recurrent disc herniation will be monitored through MRI scans and clinical evaluations. The rate of recurrence in both the FELD and MD groups will be compared to determine if one technique results in a higher recurrence rate.
Time to Return to Work | Up to 12 months post-surgery
  This measure will assess the number of days taken for patients to return to their regular work activities post-surgery, comparing the recovery times between the FELD and MD groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kajetan Latka, PhD, Principal Investigator — University of Opole
Locations (2):
- Poland (2):
  - Uniwesytecki Szpital Kliniczny, Opole, Opole Voivodeship
  - Wojewódzki Szpital Specjalistyczny im Św Jadwigi w Opolu, Opole, Opole Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
The following specific Individual Participant Data (IPD) will be shared:
  * De-identified individual clinical data: This includes data from questionnaires such as Visual Analog Scale (VAS), Core Outcome Measures Index (COMI), and Oswestry Disability Index (ODI), collected at baseline and during follow-up visits (1, 3, 6, and 12 months post-surgery).
  * De-identified radiological data: MRI images taken 24 hours before surgery, 24 hours after surgery, and at each follow-up visit will be shared for the purpose of comparing radiological outcomes.
  * De-identified recurrence and complication data: This includes any clinical or radiological evidence of recurrent disc herniation or complications (e.g., infection, reoperation).
  The data will be made available upon reasonable request for research purposes to qualified researchers following the publication of the primary study results.